CLINICAL TRIAL: NCT01513252
Title: A 2-years Extension Study of MAPT Trial : Evaluation of the Long Term Effects of Interventional Strategies to Prevent the Decline in Cognitive Functioning in Frail Older Adults
Brief Title: Long-term Effects of Interventional Strategies to Prevent Cognitive Decline in Elderly.
Acronym: MAPT-PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/11/231; 2011-A00764-37 (Other: ID-RCB)
Record Dates: First submitted 2011-12-30; First posted 2012-01-20 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Frail Elderly
Keywords: Cognitive decline; prevention; omega-3 fatty acids; nutrition exercise; cognitive training; social activities; frailty
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Gröber and Buschke test
  Interventions: Behavioral: Gröber and Buschke test

INTERVENTIONS:
Behavioral: Gröber and Buschke test — spontaneous delayed recall score after a 5 years follow-up

SUMMARY:
The MAPT PLUS study is a two-year extension of follow-up of the patients included in the MAPT preventive study, after completion of the interventions. Subjects in the four groups of the MAPT study will be prospectively followed. MAPT is a multicentre, randomised, placebo-controlled study, using a 4-group design with 3 treatment groups (omega 3 alone, multi-domain intervention alone, omega 3 plus multi-domain intervention, n=420 each) and a placebo group (n=420). The MAPT PLUS study will be an extension of the MAPT study and includes an annual follow-up for two years.

DETAILED DESCRIPTION:
The MAPT PLUS study is a follow-up of subjects initially included in an interventional study. The follow-up that we propose in this request for funding does not involve any intervention, but aims to assess the long-term effect of the interventions previously carried out during the three years of the MAPT study.

* Description of the interventions to which subjects are exposed during the first 3 years of follow-up (MAPT study) :

In the MAPT study, subjects are randomized into 4 groups:

* V0137 CA group: 2 soft capsules of V0137 CA once a day (2 x 400 mg/day);
* Multi-domain intervention group (nutrition, physical activity, cognitive stimulation, social activities) + placebo, 2 soft capsules once a day ;
* Multi-domain intervention group (nutrition, physical activity, cognitive stimulation, social activities) + V0137 CA, 2 soft capsules once a day ;
* Placebo group: 2 soft capsules of placebo once a day. * Description of the multidomain intervention : The multi-domain intervention consists of collective training sessions and a yearly personalized preventive consultation which aims to detect risk factors (sensory disturbances, difficulty in walking, nutritional disturbances, vascular risk factors) and to set up management in collaboration with the general practitioner.

The collective sessions take place in groups of 6 to 8 subjects. In the first month, two sessions a week are scheduled, and in the second month, one session a week. The first two months correspond to the intensive programme. Each session comprises 1 hour of cognitive training, 45 minutes of information on physical activity and 15 minutes of dietary advice. From the third month, sessions are held monthly and aim to consolidate the key messages and to stimulate adherence to the programme. The sessions are shorter (1 hour review of one of the domains of the intensive programme). " Booster " sessions (2 hours) are delivered at 12 and 24 months after the first sessions of the intensive programme. Twenty-minute individual interviews also take place every 6 months with the leader of the training sessions (6 interviews in the course of 3 years).

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria will be included in the MAPT PLUS study :

* frail elderly subjects participating in the MAPT study and still followed at 3 years,
* subjects capable of understanding the protocol, complying with its requirements and attending the follow-up visits proposed as part of the extended phase of the MAPT study,
* subjects capable of giving their written informed consent and complying with the requirements of the study,
* subjects covered by a health insurance system.

Exclusion Criteria:

Subjects who fulfill at least one of the following criteria will not be included in the MAPT PLUS study :

* known presence of dementia or Alzheimer's disease (DSM IV criteria) diagnosed during the MAPT follow-up,
* known presence of severe diseases that are life-threatening in the short term,
* visual or hearing impairments that are incompatible with performance and/or interpretation of the neuropsychological tests,
* history and/or presence of any disorder (severe depression or generalized anxiety) which, according to the investigator, is likely to interfere with the results of the study or to expose the subject to a supplementary risk,
* participation in another clinical study during the period of the present study,
* subjects who have refused cognitive evaluation during the MAPT follow-up,
* subjects deprived of their freedom by administrative or judicial decision, or under guardianship,
* with regard to performance of MRI: presence of a pacemaker or metallic materials, claustrophobia.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Gröber and Buschke test (spontaneous delayed recall score) | 2 years
  Assessment of cognitive and functional performances according to the spontaneous delayed recall score(Gröber and Buschke test)
Cognitive and functional performance (Gröber and Buschke test-spontaneous delayed recall score) | 2 years
  Assessment of cognitive and functional performances by using the Gröber and Buschke test (spontaneous delayed recall score)at 5 years after the participation to the MAPT study.

SECONDARY OUTCOMES:
MRI test | 2 years
  Evaluation of the long-term impact of MAPT study interventions on changes in markers of cerebral atrophy (overall brain volume of specific brain structures such as the hippocampus)
Cost-effectiveness Evaluation | 2 years
  Evaluation of the long-term impact of the MAPT interventions in terms of cost-effectiveness ratio by using a medico-economic data collection

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vellas, MD, Principal Investigator — University Hospital, Toulouse
Locations (13):
- France (12):
  - Bordeaux, Bordeaux
  - CH Castres-Mazamet, Castres
  - CHRU Dijon, Dijon
  - CHIVA, Foix
  - LAVAUR, Lavaur
  - CHU Limoges, Limoges
  - Lyon-Sud Hospital, Lyon
  - Chg Montauban, Montauban
  - CHU Montpellier, Montpellier
  - Nice, Nice
  - Tarbes, Tarbes
  - UH Toulouse - La Grave, Toulouse
- CH Princesse Grâce, Monaco, Monaco

REFERENCES:
- [Derived] Delrieu J, Vellas B, Guyonnet S, Cantet C, Ovod V, Li Y, Bollinger J, Bateman R, Andrieu S; MAPT/DSA group. Cognitive impact of multidomain intervention and omega 3 according to blood Abeta42/40 ratio: a subgroup analysis from the randomized MAPT trial. Alzheimers Res Ther. 2023 Oct 23;15(1):183. doi: 10.1186/s13195-023-01325-3. PMID 37872582
- [Derived] Takano E, Maltais M, Kondo I, Rolland Y; MAPT/DSA group. Bidirectional relationship between depressive symptoms and physical performance in community-dwelling older people with subjective memory complaints. Eur Geriatr Med. 2021 Oct;12(5):973-980. doi: 10.1007/s41999-021-00473-9. Epub 2021 Mar 5. PMID 33666880
- [Derived] Delrieu J, Voisin T, Saint-Aubert L, Carrie I, Cantet C, Vellas B, Payoux P, Andrieu S. The impact of a multi-domain intervention on cerebral glucose metabolism: analysis from the randomized ancillary FDG PET MAPT trial. Alzheimers Res Ther. 2020 Oct 19;12(1):134. doi: 10.1186/s13195-020-00683-6. PMID 33076983
- [Derived] Delrieu J, Payoux P, Carrie I, Cantet C, Weiner M, Vellas B, Andrieu S. Multidomain intervention and/or omega-3 in nondemented elderly subjects according to amyloid status. Alzheimers Dement. 2019 Nov;15(11):1392-1401. doi: 10.1016/j.jalz.2019.07.008. Epub 2019 Sep 23. PMID 31558366
- [Derived] Pothier K, de Souto Barreto P, Maltais M, Rolland Y, Vellas B. Shifting from Declines to Improvements: Associations between a Meaningful Walking Speed Change and Cognitive Evolution over Three Years in Older Adults. J Nutr Health Aging. 2018;22(10):1183-1188. doi: 10.1007/s12603-018-1059-8. PMID 30498824
- [Derived] Lilamand M, Cesari M, Cantet C, Payoux P, Andrieu S, Vellas B; the MAPT/DSA study group. Relationship Between Brain Amyloid Deposition and Instrumental Activities of Daily Living in Older Adults: A Longitudinal Study from the Multidomain Alzheimer Prevention Trial. J Am Geriatr Soc. 2018 Oct;66(10):1940-1947. doi: 10.1111/jgs.15497. Epub 2018 Sep 12. PMID 30207586